CLINICAL TRIAL: NCT06766994
Title: The Effect of Two Different Analgesic Techniques on Postoperative Recovery Quality in Patients Undergoing Elective Abdominal Hysterectomy
Brief Title: The Effect of Two Different Analgesic Techniques on Postoperative Recovery Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Berivan Bozan, Research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: B.30.2.YYU.0.01.00.00/105
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Hysterectomy
Keywords: abdominal hysterectomy; intrathecal morphine; erector spinal plane block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intrathecal morphine (Active Comparator)
  Interventions: Other: intrathecal morphine
- Group Erector Spinae Plane Block (Active Comparator)
  Interventions: Other: Erector Spinae Plane Block

INTERVENTIONS:
Other: intrathecal morphine — Preoperatively, patients will be injected with 200 μg morphine intrathecally with a 27G pencil point spinal needle at the L4-L5 or L3-L4 intervertebral space in a sitting position.
  Arms: Group Intrathecal morphine
Other: Erector Spinae Plane Block — Preoperatively, patients will be placed in the prone position before the operation and an ESPB block will be applied bilaterally at the T9 vertebra level with the help of USG. 0.25% bupivacaine 20 ml will be used bilaterally as the blocking fluid.
  Arms: Group Erector Spinae Plane Block

SUMMARY:
Hysterectomy is one of the most frequently performed surgical procedures after Caesarean section in many countries of the world and involves the removal of the uterine corpus with or without the cervix (total hysterectomy) or without the cervix (subtotal or supracervical hysterectomy) to treat a range of gynecological problems. Hysterectomy is performed abdominally, vaginally with laparotomy, or using minimally invasive techniques (laparoscopy, robotic surgery). The abdominal route for hysterectomy is the preferred route in 60-80% of these surgeries.

Postoperative recovery is a complex condition affected by various factors such as patient characteristics, surgical procedure, and anesthesia. There are many tools available to measure recovery quality. In recent years, the concept of recovery quality perceived by the patient has attracted attention. The Quality of Recovery-40 questionnaire (QoR-40) is an assessment test used to assess recovery quality and health status in the early postoperative stages. QoR-40 consists of 40 questions that evaluate patients' pain, physical comfort, physical independence, psychological support, and emotional state. Quality of Recovery-15 (QoR-15) is a short postoperative recovery scale developed and validated by Stark et al. in 2013. It is an abbreviated version of the QoR-40 scale. It is easy to use because it is shorter and can be completed in a short time. As in QoR-40, it contains 15 questions that evaluate pain, physical comfort, physical independence, psychological support, and emotional state by the patient.

Facilitating the recovery process and optimizing postoperative pain management is an important part of perioperative care. Multimodal analgesia, which combines local anesthesia, peripheral and non-opioid analgesics to minimize systemic opioid requirements and opioid-related side effects, has become increasingly popular. Epidural analgesia, which provides both intraoperative and postoperative analgesia as a complement to general anesthesia for elective abdominal hysterectomy, is an approach applied to achieve balanced and multimodal analgesia. Thus, while the adverse effects of high doses, especially opioid analgesics, applied with a single method are reduced, more effective treatment can be provided for postoperative pain where drugs and other methods alone are insufficient to provide complete analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo abdominal hysterectomy surgery under general anesthesia
* Ages between 18-65
* American Society of Anesthesiologists classification I-II

Exclusion Criteria:

* Patients with a BMI ≥ 35,
* Patients with allergies to the drugs to be used in the study,
* Patients with severe liver or kidney failure,
* Patients with a history of long-term use of nonsteroidal anti-inflammatory and opioid analgesics,
* Patients with a history of gastrointestinal bleeding, peptic ulcers or inflammatory bowel disease,
* Patients with a history of diabetes or other neuropathic diseases,
* Patients who developed atrioventricular block and bradycardia before surgery,
* Patients with a history of serious underlying respiratory disease and psychiatric diseases,
* Patients with ASA stage 3 or higher,
* Patients who cannot use a patient-controlled analgesia (PCA) device,
* Patients who need to stop the drug used in the study during surgery for any reason,
* Patients who do not consent to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery 24 hours after surgery assessed using the QoR-15 questionnaire | postoperative 24 hours
  The primary objective of this study was to evaluate the quality of recovery 24 hours after surgery using the QoR-15 questionnaire after preoperative erector spinae plane block and intrathecal morphine injection in patients undergoing elective abdominal hysterectomy.

SECONDARY OUTCOMES:
Total amount of opioids consumed | postoperative 24 hours
  The secondary objective was to measure the total amount of opioid consumed in the first 24 hours postoperatively.
pain scores with movement and at rest | postoperative 24 hours
  Evaluation of pain scores during movement and rest within 24 hours postoperatively using the Visual Analog Scale
irst analgesic requirement | postoperative 24 hours
  Time to first analgesic requirement in the postoperative period
Advers events | postoperative 24 hours
  incidence of side effects (nausea, vomiting, pruritus, urinary retention) for 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Hein A, Rosblad P, Gillis-Haegerstrand C, Schedvins K, Jakobsson J, Dahlgren G. Low dose intrathecal morphine effects on post-hysterectomy pain: a randomized placebo-controlled study. Acta Anaesthesiol Scand. 2012 Jan;56(1):102-9. doi: 10.1111/j.1399-6576.2011.02574.x. PMID 22150410